CLINICAL TRIAL: NCT06558006
Title: Safety and Efficacy of Predimenol for Headache: A Preliminary Study
Brief Title: Safety and Efficacy Predimenol for Headache
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Collaborators: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRSU.P.Dexa/06/20/13.04
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Headache
Keywords: Predimenol; Headache
MeSH Terms: conditions — Headache

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Group (Experimental): 2 tablets of Predimenol (400 mg Predimenol)
  Interventions: Drug: Predimenol tablet
- Treatment + Placebo Group (Experimental): 1 tablet of Predimenol (200 mg Predimenol) + 1 tablet of placebo
  Interventions: Drug: Predimenol tablet + Placebo tablet of Predimenol
- Control Group (Placebo Comparator): 2 tablets of placebo
  Interventions: Drug: Placebo tablet of Predimenol

INTERVENTIONS:
Drug: Predimenol tablet — 2 tablets of Predimenol (400 mg Predimenol) will be taken with 220 mL of water (one glass of water).
  Other Names: HerbaPAIN
  Arms: Treatment Group
Drug: Predimenol tablet + Placebo tablet of Predimenol — 1 tablet of Predimenol (200 mg Predimenol) + 1 tablet of placebo will be taken with 220 mL of water (one glass of water).
  Arms: Treatment + Placebo Group
Drug: Placebo tablet of Predimenol — 2 tablets of placebo tablet of Predimenol will be taken with 220 mL of water (one glass of water).
  Arms: Control Group

SUMMARY:
This is a prospective, double-blind, placebo-controlled and randomized study aimed to obtain a description of the efficacy and safety of Predimenol in alleviating headache.

DETAILED DESCRIPTION:
Predimenol is a bioactive fraction extracted from Phaleria macrocarpa pericarpium (Mahkota Dewa).

There will be 20 subjects per group (a total of 60 subjects) planned to be enrolled in the study.

The investigational drug: tablet @200 mg of Predimenol. Dose administration: one singe dose (two tablets) of Predimenol or Placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men or women aged 18 to 60 years with acute moderate tomoderate-severe headache.
2. Signing the informed consent.

Exclusion Criteria:

1. Body temperature of >37.3˚C and/or refuse to follow health protocol for COVID-19.
2. Known hypersensitivity to herbal drugs.
3. Pregnant or lactating women.
4. Have received any analgesic or anti-inflammatory drugs within the past 12 hours.
5. Presence of vomiting or diarrhea within the past 24 hours or still ongoing at the start of study.
6. Severe illness, e.g. severe hypertension, or any known organic diseases that may cause headache.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-19 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Time 0, 10 min, 20 min, 30 min, 1 hour, 2 hour
  VAS (Visual Analogue Scale) for headache (0 - 100), with 0 indicates asymptomatic and 100 refers to the most serious or severe symptom.
  VAS will be measured at baseline and 10 min, 20 min, 30 min, 1 hour, 2 hour after drug administration.
Adverse events | Time 0, 10 min, 20 min, 30 min, 1 hour, 2 hour
  Any kind of adverse events (AE) and serious adverse events (SAE) will be observed throughout the study conduct.

CONTACTS AND LOCATIONS:
Overall Officials: Nalfriadi Nalfriadi, MD,SpPD,PhD, Principal Investigator — Department Pharmacology & Therapeutics Faculty of Medicine Universitas Indonesia
Locations (2):
- Indonesia (2):
  - Imeri Fkui, Jakarta Pusat, DKI Jakarta
  - Klinik Satelit Makara UI Depok, Depok, West Java